CLINICAL TRIAL: NCT05715008
Title: The Effect of Kefir Consumption on Anthropometric, Physiological and Oxidative Stress Parameters in Adults Subjects
Brief Title: Kefir Consumption on Various Parameters in Adults Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTH_Kefir
Record Dates: First submitted 2023-01-07; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — Kefir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kefir consumption (Experimental): Kefir consumption (300ml/day) for 2 weeks in a counterbalanced manner to 16 adult subjects
  Interventions: Other: Kefir
- Placebo (cow milk) (Placebo Comparator): Placebo administration for 2 weeks in a counterbalanced manner to 16 adult subjects
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Kefir — Comparison of kefir and placebo consumption for 2 weeks on various parameters in healthy adult subjects
  Arms: Kefir consumption
Other: Placebo — Comparison of kefir and placebo consumption for 2 weeks on various parameters in healthy adult subjects
  Arms: Placebo (cow milk)

SUMMARY:
The purpose of this study is to examine the effect of kefir consumption on anthropometric, physiological and redox status parameters in adult subjects, and compare it with the intake of placebo drink (milk).

DETAILED DESCRIPTION:
Importance of the research

Several chronic diseases are related with alterations in redox status. Over the years several nutritional approaches have been implemented in order to examine modulation of the redox status. Kefir is a product that can alter the gut microbiome and potentially affect the redox status. This study will help elucidate whether the consumption of a dairy product (kefir) will modulate anthropometric, physiological and oxidative stress parameters.

Methodology

1. Sample:

   The study will involve 16 adult volunteers, (8-experimental group and 8-control group), aged 20-60 years. The subjects will participate in a double-blind, randomized study, where in one condition they will receive kefir (300 ml per day - 150 ml in the morning and 150 ml in the evening) and in the next condition they will receive regular cow milk as a placebo.
2. Process of collecting results:

   At first visit of volunteers to the laboratory, anthropometric (height, weight, body fat percentage, waist and hip circumferences) and physiological measurements (heart rate, blood pressure) will be taken. Volunteers will also be given full instructions on how to record their diet. They will be given a form to record their diet for 3 days and will have to follow the same date before each next visit to the laboratory.

   Then they will have their second visit to the laboratory, where the first blood sampling will be taken, and they will be given the necessary amount of kefir or placebo (depending on the group to which they belong), which they will have to consume as a supplement for the following two weeks.

   At the end of the 2 weeks the volunteer will return to the laboratory where the second blood sampling will be performed.

   This will be followed by a 2-week washout period where participants will not receive any amount of kefir or placebo. At the end of this intervention, a fourth visit to the laboratory will take place, where the third blood sampling will be performed.

   Subsequently, the consumption of kefir or placebo will continue, except that participants who initially consumed kefir will receive the placebo and vice versa.

   The last blood sampling (fourth) will take place after two weeks.
3. Measuring instruments:

   Dual-energy X-ray absorptiometry (DEXA) and a mechanical balance with a stadiometer will be used to determine the anthropometric characteristics.

   A Gulick tape measure will be used to measure the waist and hip circumferences.

   For the measurement of heart rate a polar type heart rate monitor will be used.

   A sphygmomanometer will be used to measure blood pressure.

   The dietary characteristics of their diet will be analysed using a Science Fit Diet 200A (ScienceFit, Greece).

   Parameters in the blood will be analyzed by Immunoenzymatic Analysis (ELISA) and visible-ultraviolet spectrophotometer.
4. Blood parameters:

A portion of the blood will be utilized for a complete blood count analysis and parameters related to redox status (protein carbonyls, thiobarbituric acid reactive substances, reduced glutathione, oxidized glutathione, catalase, total antioxidant capacity, uric acid).

Statistical Analysis

A 2-way ANOVA with repeated measures will be performed. The statistical program SPSS 26 will be used.

ELIGIBILITY:
Inclusion Criteria:

* The persons selected will be volunteers.
* The use of alcohol and smoking will be prohibited during the experiment.
* Participation in other sports activities will also not be allowed.
* In the last six months they should not have taken any medication that affect the redox status, as well as dietary supplements with antioxidants.
* Their blood pressure should be within normal limits.

Exclusion Criteria:

* Individuals with a past of health problems that are likely to have a negative effect on the indicators to be tested.
* Individuals with allergies.
* People with liver and gastric tract problems (e.g. ulcers).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Changes in total antioxidant capacity following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using 2,2-diphenyl-1-picrylhydrazyl (DPPH) method.
Changes in glutathione following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using 5,5'-dithio-bis-(2-nitrobenzoic acid) (DTNB) method.
Changes in uric acid following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using a clinical chemistry analyzer with commercially available kits.
Changes in bilirubin following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Index of blood redox status. Spectrophotometric assay for the determination of bilirubin using a clinical chemistry analyzer with commercially available kits.
Changes in lipid peroxidation following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Index of blood redox status. Determination of lipid peroxidation using malondialdehyde production assessment.
Changes in protein carbonyls following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using 2,4-Dinitrophenylhydrazine (DNPH) method.

SECONDARY OUTCOMES:
Changes in body composition (in kg) following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Body mass (in kg), body fat mass (in kg), lean mass (in kg)
% Changes in body composition following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Body fat mass percentage, lean mass percentage
Changes in body mass index following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Body mass (in kg) and height (in cm).
Changes in waist-to-hip ratio following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Measurement of waist and hip circumference to calculate waist-to-hip ratio.
Changes in blood pressure following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Measurement of (systolic and diastolic) blood pressure (in mm Hg) after at least 5 minutes at rest.
Changes in resting heart rate following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Resting heart rate (beats per minute) measurement after at least 5 minutes at rest.
Changes in red blood count (RBC) following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  RBC (million cells per microliter)
Changes in hemoglobin (HGB) following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  HGB (grams per deciliter)
Changes in hematocrit (HCT), Red blood cell Distribution Width (RDW), Plateletcrit (PCT) and Platelet Distribution Width (PDW) following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  HCT (%), RDW (%), PCT (%), PDW (%)
Changes in Mean Corpuscular Volume (MCV) and Mean Platelet Volume (MPV) following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  MCV and MPV (fL)
Changes in Mean Corpuscular Hemoglobin (MCH) following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  MCH (pg)
Changes in Platelets, White Blood Cell Count (WBC), Neutrophils, Granulocytes, Monocytes following 2 weeks of kefir consumption and placebo. | 2 weeks (Before and after 2 weeks of kefir consumption and before and after 2 weeks of placebo).
  Platelets, WBC, Neutrophils, Granulocytes and Monocytes (in thousand cells per microliter)

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, PhD, Study Director — University of Thessaly